CLINICAL TRIAL: NCT01492881
Title: A Multi-Center, Single-Arm, Phase II Study of Vorinostat (V) in Combination With Pegylated Liposomal Doxorubicin (PLD) and Bortezomib (B) Followed by VB Maintenance in Patients With Relapsed and Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Vorinostat With Doxil and Bortezomib for Patients With Relapsed/Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Doxil is currently unavailable
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1119
Record Dates: First submitted 2011-12-12; First posted 2011-12-15 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Myeloma
Keywords: relapsed multiple myeloma; refractory multiple myeloma; vorinostat; bortezomib; doxil
MeSH Terms: conditions — Multiple Myeloma | interventions — Vorinostat; Bortezomib; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat, Bortezomib, Doxil (Experimental): Induction therapy will consist of up to 8 cycles of vorinostat, bortezomib, and doxil. One cycle is defined as 21 days.
  Maintenance therapy will consist of Vorinostat and bortezomib. One maintenance cycle is 28 days and repeated for up to 1 year.
  Interventions: Drug: Vorinostat; Drug: Bortezomib; Drug: pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: Vorinostat — Oral, 400mg, taken days 4 through 11 of each cycle.
  Other Names: Zolina
Drug: Bortezomib — subcutaneous injection, 1.3mg/m2, Days 1, 4, 8, and 11 every cycle
  Other Names: Velcade
Drug: pegylated liposomal doxorubicin — Intravenous, 30mg/m2, Day 4
  Other Names: Doxil

SUMMARY:
The purpose of this research study is to determine how multiple myeloma responds when the study drug vorinostat is added to the standard treatment of bortezomib and pegylated liposomal doxorubicin (PLD). After participants complete the three drug combination and if their multiple myeloma has decreased, the investigators also want to learn what effects (both good and bad) when vorinostat and bortezomib are given to people with multiple myeloma over a longer period of time. This type of treatment is called 'Maintenance Therapy'.

DETAILED DESCRIPTION:
This is a prospective, open-label single arm phase II trial of vorinostat, bortezomib and pegylated liposomal doxorubicin (PLD) followed by vorinostat/bortezomib (VB) maintenance therapy for patients with relapsed and relapsed and refractory multiple myeloma (MM). The primary hypothesis being evaluated is that the addition of vorinostat to the PLD and bortezomib backbone (VB-PLD) will improve the overall response rate (ORR) as compared to a historical control of PLD in combination with bortezomib.[1] We anticipate that the addition of maintenance therapy will not improve the ORR, but may improve the quality (depth) of response and progression free survival (PFS).

Secondary endpoints include PFS, high quality response rates (very good partial responses (VGPR) + complete responses (CRs)), duration of remission (DOR), quality of life (QOL), overall survival (OS) and tolerability of the regimen in patients with relapsed and relapsed and refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

Relapsed or relapsed and refractory multiple myeloma:

* Relapsed MM is defined as clinically active disease, in patients who have received one or more prior therapies, that is not refractory to the most recent treatment. (Refractory to the prior treatment means either progressive disease (PD) on last prior therapy; best response of stable disease (SD) to last prior therapy, or PD within 60 days of completing therapy).
* Relapsed and refractory MM is defined as relapsed disease, which either becomes non-responsive while on salvage therapy, or progresses within 60 days of last therapy.

  1 to 3 prior lines of therapy for multiple myeloma (a single line of treatment may consist of 1 or more agents and regimens. A single line of therapy may be most easily delineated by a response to treatment followed by a change in treatment due to the progression of disease.
* Prior bortezomib- and anthracycline-based therapy is allowed; prior cumulative doxorubicin dose must be <360 mg/m2 (or its equivalent)
* Prior autologous stem cell transplantation is allowed provided the patient is 3 months out from transplant and has recovered from any transplant-related toxicities (to baseline or grade 1 in severity)

All prior treatment-related non-hematologic toxicities resolved to ≤Grade 1 (or baseline), not including alopecia

Prior radiation therapy completed ≥2 weeks prior to day 1 of treatment Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Age ≥18 years

Life expectancy of at least 6 months

Adequate bone marrow function (without platelet or RBC transfusion support within one week of screening) as demonstrated by:

* Hemoglobin ≥ 8 g/dL (use of erythropoietin stimulating agent is OK)
* Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3 (without granulocyte growth factor support)
* Platelet count ≥ 100,000/mm3 (≥75,000/mm3 in patients with ≥30% marrow involvement of MM who are felt to have thrombocytopenia primarily due to marrow infiltration of disease as opposed to diminished marrow reserves from prior therapy)

Adequate hepatic and renal function as demonstrated by:

* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
* Total serum bilirubin ≤1.5 x ULN
* Creatinine clearance (CrCL) ≥ 30mL/min as measured via Cockcroft-Gault or 24-hour urine testing

Documented negative serologic testing for hepatitis B (HBV) and Hepatitis C (HCV) as measured by the following (NOTE: this testing is not necessary if patient has had negative testing within the last year, and no subsequent risk factors for acquisition of these viruses):

* HBV surface antigen, surface antibody, and core antibody (NOTE: patients who are seropositive because of hepatitis B vaccine are eligible)
* HCV antibody.
* For patients with serologic evidence of viral hepatitis, quantitative PCR will be performed.

Documented negative HIV blood test (NOTE: this testing is not necessary if patient has had negative testing within the last year, and no subsequent risk factors for acquisition of this virus)

Adequate cardiac function, defined as:

* No EKG evidence of acute ischemia
* No EKG evidence of active clinically significant conduction system abnormalities
* No EKG evidence of > Grade 2 (>480 ms) QTc prolongation
* Prior to study entry, any ECG abnormality at screening not felt to put the patient at risk has to be documented by the investigator as not medically significant
* No uncontrolled angina or severe ventricular arrhythmias
* No clinically significant pericardial disease
* No history of myocardial infarction within the last 6 months
* Left ventricular ejection fraction (LVEF) must be > 45% by either echocardiography or radionuclide-based multiple gated acquisition (MUGA)
* No Class II or higher New York Heart Association Congestive Heart Failure

Negative serum β-hCG pregnancy test within 72 hours of day 1 of treatment with study medications in women of child-bearing potential

All males and females of childbearing potential must agree to use an effective contraceptive method during the study and for 3 months following the last dose of study treatment. Effective contraception is defined as any medically recommended method (or combination of methods) as per standard of care, including abstinence. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy

Exclusion Criteria:

* > 3 prior lines of therapy for treatment of MM

Receipt of prior allogeneic stem cell/bone marrow transplantation

Primary refractory MM as defined by the ASH/FDA Workshop on Clinical Endpoints in Multiple Myeloma[24]

Peripheral neuropathy (PN) ≥ grade 1 with pain or ≥grade 2 PN within 14 days prior to enrollment

Known history of HIV, HBV or HCV infection

Serum potassium ≤3.0 mmol/L or serum magnesium ≤1.6mg/dL that cannot be corrected with supplementation

Known hypersensitivity to bortezomib or any of its components (boron, mannitol), vorinostat, doxorubicin, or any of the components of PLD; Patients with a history of reactions to other liposomal drug formulations will be evaluated individually, and if their reactions were felt to have been due to the liposome itself, as opposed to the encapsulated agent, they will be excluded at the discretion of the investigators.

Prior or concomitant use of a histone deacetylase inhibitor (exception: prior valproic acid for epilepsy is allowed provided patient undergoes a 30 day wash out prior to D1 of study treatment)

No major surgery within 3 weeks prior to day 1 of study treatment

Active, serious infection, medical, or psychiatric condition that would represent an inappropriate risk to the patient or would likely compromise achievement of the primary study objective

Other prior or concomitant malignancies with the exception of:

* Non-melanoma skin cancer
* In-situ malignancy
* Low-risk prostate cancer after curative therapy
* Other cancer for which the patient has been disease free for ≥ 3 years

Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Estimate the overall response rate. | 18 months
  Estimate the overall response rate (ORR) of the vorinostat, PLD and bortezomib regimen (VB/PLD) followed by vorinostat/bortezomib (VB) maintenance in patients with relapsed and relapsed/refractory multiple myeloma. Criteria for response will be based on the International Uniform Response Criteria for Multiple Myeloma, modified to incorporate criteria for minor response (MR). The overall response rate will be defined as the total number of patients whose response are PR or above, divided by the number of response evaluable patients.

SECONDARY OUTCOMES:
Evaluate the quality of life measures in patients. | 18 months
  QOL will be evaluated using the EORTC QLQ-C30 and QLQ-MY20 survey instruments.
Assess the safety and tolerability. | 18 months
  Safety will be assessed via the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4 (CTCAE v4). The analysis of safety will be based on the frequency of adverse events and their severity for patients who received any study medicine.
Estimate the overall survival. | 36 months
  A patient's survival time will be defined as the time from start of treatment to the date of his or her death.
Estimate Progression-free survival | 36 months
  A patient's progression-free survival (PFS) will be defined as the time from start of treatment until the date he or she has documented progression or dies.

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Voorhees, MD, Principal Investigator — Lineberger Comprehensive Cancer Center at University of North Carolina at Chapel Hill
Locations (1):
- Lineberger Comphrehensive Cancer Center at University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center N.C. Cancer Hospital — http://unclineberger.org/